CLINICAL TRIAL: NCT01183468
Title: Effect of Intravenous Alpha-1 Antitrypsin on Preserving Beta-cell Function in New-onset Type 1 Diabetes Mellitus (ITN041AI)
Brief Title: A Research Trial of Aralast in New Onset Diabetes (RETAIN)
Acronym: RETAIN
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to lack of mechanistic signal and competing industry studies
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN041AI Part 1
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1 (new-onset); Diabetes Mellitus, Insulin-Dependent (new-onset); new-onset T1DM; new-onset T1D; Diabetes Mellitus, Juvenile-Onset; Diabetes, Autoimmune; Aralast NP; Alpha-1 Antitrypsin; AAT
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1a(Aralast NP)-Subjects Aged 16-35 Yrs (Experimental): Subjects aged 16-35 years at enrollment with new-onset type 1 diabetes mellitus (T1DM) received Aralast NP 45 mg/kg by intravenous (IV) infusion once a week for 6 weeks. Following the Week 6 infusion, participants underwent a minimum 3-week washout period. After the washout period, each participant proceeded to a high dose of Aralast NP 90 mg/kg by IV infusion for the next 6 weeks, for a total of 12 infusions.
  Interventions: Biological: Aralast NP 45 mg dose; Biological: Aralast NP 90 mg dose
- Part 1a (Aralast NP)-Subjects 8-15 Yrs (Experimental): Subjects aged 8-15 years at enrollment with new-onset type 1 diabetes mellitus (T1DM) received Aralast NP 45 mg/kg by IV infusion once a week for 6 weeks. Following the Week 6 infusion, participants underwent a minimum 3-week washout period. After the washout period, each participant proceeded to a high dose of Aralast NP 90 mg/kg by IV infusion for the next 6 weeks, for a total of 12 infusions.
  Interventions: Biological: Aralast NP 45 mg dose; Biological: Aralast NP 90 mg dose
- Part 1b (Aralast NP)--Subjects Aged 18-35 Yrs (Experimental): Aralast NP 90 mg/kg/wk by IV infusion once a week for 6 weeks. Following the Week 6 infusion, participants undergo a minimum 3-wk washout period than then, each participant proceeds to high dose Aralast NP 180 mg/kg/wk by IV infusion for the next 6 weeks, for a total of 12 infusions.
  Interventions: Biological: Aralast NP 90 mg dose; Biological: Aralast NP 180 mg dose
- Part 1b (Aralast NP)-Subjects 8-17 Yrs (Experimental): Aralast NP 90 mg/kg/wk by IV infusion once a week for 6 weeks. Following the Week 6 infusion, participants undergo a minimum 3-wk washout period than then, each participant proceeds to high dose Aralast NP 180 mg/kg/wk by IV infusion for the next 6 weeks, for a total of 12 infusions.
  Interventions: Biological: Aralast NP 90 mg dose; Biological: Aralast NP 180 mg dose

INTERVENTIONS:
Biological: Aralast NP 45 mg dose — - 45 mg/kg/week
  Other Names: Alpha 1-Antitrypsin; AAT
  Arms: Part 1a (Aralast NP)-Subjects 8-15 Yrs; Part 1a(Aralast NP)-Subjects Aged 16-35 Yrs
Biological: Aralast NP 90 mg dose — - 90 mg/kg/week
  Other Names: Alpha 1-Antitrypsin; AAT
Biological: Aralast NP 180 mg dose — - 180 mg/kg/week
  Other Names: Alpha-1 Antitrypsin; AAT
  Arms: Part 1b (Aralast NP)--Subjects Aged 18-35 Yrs; Part 1b (Aralast NP)-Subjects 8-17 Yrs

SUMMARY:
The drug Alpha-1 Antitrypsin (AAT, Aralast NP) is being tested in this study as an anti-inflammatory drug (a medication that decreases inflammation, which is part of the body's normal ability to fight infection and respond to injuries) that affects the cells thought to be involved in the development of type 1 diabetes mellitus (T1DM, T1D).

All subjects enrolled in this study have new-onset T1DM (diagnosis of T1DM within 100 days of Visit 0; T1DM diagnosis fulfilling American Diabetes Association standard T1DM criteria). The focus of Part I of this trial (NCT01183468) is pharmacokinetics (PK), pharmacodynamics (PD) and safety. Upon completion of Part I, including a satisfactory safety review, enrollment in Part II (NCT01183455, Phase II Clinical Trial) will begin.

DETAILED DESCRIPTION:
Researchers are interested in conducting this study to assess whether Aralast NP (AAT, Alpha-1 Antitrypsin ) will help slow the progression of T1DM.

Part I of this study has two parts:-1a and -1b:

Part 1a (Complete): An open-label, dose-escalation, PK, PD and safety study. Participants receive 12 intravenous (IV) infusions of Aralast NP. Infusions 1 through 6 are administered at 45 mg/kg/wk and infusions 7 through 12 are administered at 90 mg/kg/wk.

Part Ia consists of two groups:

* Subjects aged 16 - 35 years at enrollment with new-onset T1DM
* Subjects aged 8 -15 years at enrollment with new-onset T1DM.

Part 1b (study terminated prior to subject enrollment): An open-label, dose-escalation PK, PD and safety study in which participants receive 12 infusions of Aralast NP. Infusions 1 through 6 are administered at 90 mg/kg/wk and infusions 7 through 12 are administered at 180 mg/kg/wk. Part Ib consists of two groups:

* Subjects aged 16 - 35 years at enrollment with new-onset T1DM
* Subjects 8 - 15 years at enrollment with new-onset T1DM.

Participants in Part Ib do not roll over into Part II (Refer to NCT01183455).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T1DM within the past 100 days (of enrollment)
* Positive for at least one diabetes-related autoantibody (Anti-GAD; Anti-insulin, if obtained within 10 days of the onset of insulin therapy; IA-2 antibody and/or ICA, or ZnT8.)
* Peak stimulated C-peptide level > 0.2 pmol/mL following a mixed meal tolerance test (MMTT)

Exclusion Criteria:

* Severe active disease (chronic active hepatitis; cardiac, pulmonary disease, hepatic, renal or immunodeficiency)
* History of any bleeding or clotting factor deficiencies, or stroke
* History of vascular disease or significant vascular abnormalities
* Positive serology of exposure to (hepatitis B virus) HBV, HCV (hepatitis C virus), HIV (human immunodeficiency virus) or toxoplasmosis
* Clinically active infection with EBV (Epstein-Barr virus), CMV (cytomegalovirus), or tuberculosis(TB)
* Prior or current use of oral, inhaled or intranasal glucocorticoids, or any medication known to cause a significant, ongoing change in the course of T1DM or immunologic status
* Prior treatment with Alpha 1-Antitrypsin (Aralast NP, AAT) or hypersensitivity to alpha 1-antitrypsin or human plasma-derived products
* Current or prior (within the last 30 days) use of metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin
* Current use of any medication known to influence glucose tolerance (e.g., beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine anti-malarial drugs, lithium, niacin)
* Females who are pregnant or lactating, or are unwilling to defer pregnancy during study participation
* IgA (immunoglobulin A) deficiency
* Uncontrolled hypertension
* Current life-threatening malignancy
* Any condition that in the investigator's opinion may compromise study participation or may confound the interpretation of the study results.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Weir, MD, Study Chair — Joslin Diabetes Center
Locations (15):
- United States (15):
  - RADY Children's Hospital (University of California, San Diego), San Diego, California
  - Barbara Davis Center (University of Colorado), Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Children's Hospital of Atlanta (Emory University), Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Naomi Berrie Diabetes Center (Columbia University), New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pacific Northwest Research Institute-University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal.
Time Frame: IPD is now available in TrialShare.
Access Criteria: Open to the public.
URL: https://www.itntrialshare.org/project/Studies/ITN041AIPUBLIC/Study%20Data/begin.view?pageId=study.DATA_ANALYSIS

REFERENCES:
- [Derived] Ozeri E, Mizrahi M, Shahaf G, Lewis EC. alpha-1 antitrypsin promotes semimature, IL-10-producing and readily migrating tolerogenic dendritic cells. J Immunol. 2012 Jul 1;189(1):146-53. doi: 10.4049/jimmunol.1101340. Epub 2012 May 25. PMID 22634621
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- See also: Juvenile Diabetes Research Foundation (JDRF) — http://jdrf.org/about-jdrf/
- Available data/document: Individual Participant Data Set: RETAIN ITN041AI — https://www.itntrialshare.org/project/Studies/ITN041AIPUBLIC/Study%20Data/begin.view?pageId=study.DATA_ANALYSIS — RETAIN ITN041AI is the Study Identifier in the Immune Tolerance Network (ITN) TrialShare Clinical Trials Research Portal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve of the fifteen centers enrolled a total of 17 newly diagnosed (within 100 days of Visit 0 first low dose infusion) Type 1 Diabetes Mellitus participants.
Groups:
- Part 1b (Aralast NP)-Subjects Aged 18-35 Yrs; Part 1b (Aralast NP)-Subjects 8-17 Yrs: Aralast NP 90 mg/kg/wk by IV infusion once a week for 6 weeks. Following the Week 6 infusion, participants undergo a minimum 3-wk washout period than then, each participant proceeds to high dose Aralast NP 180 mg/kg/wk by IV infusion for the next 6 weeks, for a total of 12 infusions.
  Aralast NP 90 mg dose: - 90 mg/kg/week
  Aralast NP 180 mg dose: - 180 mg/kg/week
Period: Overall Study
Arm/Group | Part 1a(Aralast NP)-Subjects Aged 16-35 Yrs | Part 1a (Aralast NP)-Subjects 8-15 Yrs | Part 1b (Aralast NP)-Subjects Aged 18-35 Yrs | Part 1b (Aralast NP)-Subjects 8-17 Yrs
Started | 8 | 9 | 0 | 0
Completed | 5 | 7 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1a(Aralast NP)-Subjects Aged 16-35 Yrs | Part 1a (Aralast NP)-Subjects 8-15 Yrs | Part 1b (Aralast NP)-Subjects Aged 18-35 Yrs | Part 1b (Aralast NP)-Subjects 8-17 Yrs | Total
Number analyzed (Participants) | 8 | 9 | 0 | 0 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 9 |  |  | 13
  Between 18 and 65 years | 4 | 0 |  |  | 4
  >=65 years | 0 | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.6 (5.7) | 10.7 (2.2) |  |  | 15.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 |  |  | 6
  Male | 5 | 6 |  |  | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 |  |  | 17

OUTCOME MEASURES:

1. Primary Outcome: C-peptide 2-hour AUC in Response to a Mixed-meal Tolerance Test at Week 52
Description: No results for the primary outcome measure are available since the study was terminated prior to reaching the outcome measure time frame of 52 weeks.
Time Frame: Week 52
Population: Enrolled Sample
Arm/Group | Part 1a(Aralast NP)-Subjects Aged 16-35 Yrs | Part 1a (Aralast NP)-Subjects 8-15 Yrs | Part 1b (Aralast NP)-Subjects Aged 18-35 Yrs | Part 1b (Aralast NP)-Subjects 8-17 Yrs
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2.5 years, from the start of the study in January 2011 until the last participant completed the study in July 2013.
Description: Adverse events were collected from the time a participant signed informed consent until the time an event resolved or until 30 days after the participant completed study treatment, whichever came first.
Groups:
- Subjects Aged 16 - 35 Years: Subjects aged 16-35 years at enrollment with new-onset type 1 diabetes mellitus (T1DM) received Aralast NP 45 mg/kg by IV infusion once a week for 6 weeks. Following the Week 6 infusion, participants underwent a minimum 3-week washout period. After the washout period, each participant proceeded to a high dose of Aralast NP 90 mg/kg by IV infusion for the next 6 weeks, for a total of 12 infusions.
- Subjects Aged 8 - 15 Years: Subjects aged 8-15 years at enrollment with new-onset type 1 diabetes mellitus (T1DM) received Aralast NP 45 mg/kg by IV infusion once a week for 6 weeks. Following the Week 6 infusion, participants underwent a minimum 3-week washout period. After the washout period, each participant proceeded to a high dose of Aralast NP 90 mg/kg by IV infusion for the next 6 weeks, for a total of 12 infusions.
Arm/Group | Subjects Aged 16 - 35 Years | Subjects Aged 8 - 15 Years
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/9
Other Adverse Events (participants affected / at risk) | 8/8 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Aged 16 - 35 Years (N=8) | Subjects Aged 8 - 15 Years (N=9)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Aged 16 - 35 Years (N=8) | Subjects Aged 8 - 15 Years (N=9)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (12)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5)
Chest pain (General disorders) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Infusion site haematoma (General disorders) | 0 (0) | 1 (4)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (3)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (10)
Urinary tract infection (Infections and infestations) | 2 (9) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fibrin D dimer increased (Investigations) | 0 (0) | 3 (3)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (69) | 8 (104)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 4 (77)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 2 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (9)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This (Part 1) was the drug dosing portion of the study; however, due to lack of a mechanistic signal and competing industry studies, the study was terminated and the trial portion (Part II, NCT01183455) was withdrawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No